CLINICAL TRIAL: NCT02044627
Title: A Phase 1, Open-Label,Single Radiolabeled Dose Study to Investigate the Absorption, Metabolism and Excretion of [14C]-ETC-1002 in Healthy Male Volunteers
Brief Title: Single Radiolabeled Dose Study to Investigate the Absorption, Metabolism and Excretion of [14C]-ETC-1002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1002-011
Record Dates: First submitted 2014-01-21; First posted 2014-01-24 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 dose of [14C-ETC-1002] (Experimental)
  Interventions: Drug: [14C-ETC-1002]

INTERVENTIONS:
Drug: [14C-ETC-1002]

SUMMARY:
This Phase 1 study will assess the mass balance recover of carbon-14 (14C) labelled ETC-1002 and the routes and rates of excretion of [14C]-ETC-1002

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male Volunteers
* BMI 10-35 kg/m2

Exclusion Criteria:

* Hx of CV, renal, hepatic, chronic respiratory or GI disease
* Hx of drug or alcohol abuse
* smoking within 12 mos of screening

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Level of [14C]-ETC-1002 in urine and feces after a single dose | 11 days
  using mass balance recovery

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MBChB, DRCOG, DCPSA, MFPM, Principal Investigator — Quotient Clinical, Mere Way, Ruddington Fields, Ruddington, Nottinham NG11 6JS, UK
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom